CLINICAL TRIAL: NCT02868944
Title: Interest of the Injection of Morphine, in Addition to a Local Anesthetic When Performing a Combined Spinal-epidural for Labor Analgesia
Acronym: MASEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PA14018
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Pregnant Women
MeSH Terms: interventions — Anesthetics, Local; Levobupivacaine; Morphine; Sufentanil; Single Person

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- experimental group (Experimental): sequential combined spinal epidural with local anesthetic injection associated with morphine
  Interventions: Drug: experimental group : sequential combined spinal epidural with local anesthetic injection (chirocaine) associated with morphine (sufentanil).
- control group (Active Comparator): sequential combined spinal epidural with local anesthetic injection alone
  Interventions: Drug: control group : sequential combined spinal epidural with local anesthetic injection (chirocaine) alone.

INTERVENTIONS:
Drug: experimental group : sequential combined spinal epidural with local anesthetic injection (chirocaine) associated with morphine (sufentanil).
  Arms: experimental group
Drug: control group : sequential combined spinal epidural with local anesthetic injection (chirocaine) alone.
  Arms: control group

SUMMARY:
The addition of morphine to a local anesthetic when performing an epidural analgesia during labor analgesia has improved the efficiency and the action duration of analgesia. One limitation of this technique is the time of installation of the analgesic effect (about 30 minutes) when using the only epidural. Therefore, the technique of sequential combined spinal epidural was introduced. This is to shorten the installation time by direct injection into the cerebrospinal fluid. This allows a good efficiency in less than 10 minutes. It has been shown that low doses of sufentanil (strong opioid) in spinal anesthesia could potentiate the effect of the local anesthetic.

DETAILED DESCRIPTION:
Compare the results of obstetric analgesia by sequential combined spinal epidural with local anesthetic injection associated with morphine and a sequential obstetric analgesia by sequential combined spinal epidural with local anesthetic injection alone

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients
* patients who experienced a physiological course of pregnancy
* patients for which it was estimated eutrophic fetus without pathology found during ultrasound
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years and younger than 40 years

Exclusion Criteria:

* twin pregnancy
* contraindication to sequential combined spinal epidural

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Visual analog pain scale | after 5 minutes
  Pain evaluated inferior at 3 on 10 using a visual analog pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France